CLINICAL TRIAL: NCT02381288
Title: A Randomized, Single-Blind, Placebo-Controlled Phase 2a Study to Evaluate the Stimulatory Effects of TAK-448, a Kisspeptin Analog, Administered Intermittently in Middle-aged and Older Men With Low Testosterone
Brief Title: Effects of TAK-448 in Middle-aged and Older Men With Low Testosterone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study because the study did not meet the primary endpoint.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAK-448-2002; U1111-1150-2776 (Registry Identifier: WHO)
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Low Testosterone
Keywords: Drug therapy
MeSH Terms: interventions — metastin (46-54), acetyl-tyrosyl(46)-hydroxypropyl(47)-threonyl(49)-azaglycyl(51)-methylarginyl(53)-tryptophyl(54)-

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TAK-448 0.1 mcg (Experimental): TAK-448 0.1 mcg, injection, subcutaneously, once daily on Days 1 through 42.
  Interventions: Drug: TAK-448
- TAK-448 0.3 mcg (Experimental): TAK-448 0.3 mcg, injection, subcutaneously, twice-weekly on Days 1 through 39.
  Interventions: Drug: TAK-448
- TAK-448 1.0 mcg (Experimental): TAK-448 1.0 mcg, injection, subcutaneously, once-weekly on Days 1 through 36.
  Interventions: Drug: TAK-448
- Placebo (Placebo Comparator): TAK-448 placebo matching injection, subcutaneously, either once daily on Days 1 through 42, or twice weekly on Days 1 through 39 or once weekly on Days 1 through 36.
  Interventions: Drug: TAK-448; Drug: TAK-448 Placebo

INTERVENTIONS:
Drug: TAK-448 — TAK-448 solution for subcutaneous injection
Drug: TAK-448 Placebo — TAK-448 placebo-matching solution for subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects on serum testosterone (ST) after 6 weeks of subcutaneous (SC) administration of different doses and dosing frequencies of TAK-448 to middle-aged and older men with low ST levels.

DETAILED DESCRIPTION:
The drug tested in this study is called TAK-448. TAK-448 was tested to define a dose and dose frequency which results in a clinically relevant improvement in ST in middle-aged and older men with low ST levels. This study looked at ST levels in men who took TAK-448.

The study enrolled 17 participants. Participants were randomly assigned (by chance, like flipping a coin) to one of the following treatment groups-which remained undisclosed to the participants and study doctor during the study (unless there is an urgent medical need):

* TAK-448 0.1 µg
* TAK-448 0.3 µg
* TAK-448 1.0 µg
* Placebo (dummy inactive injection) - this was a injection that looks like the study drug but has no active ingredient All participants received subcutaneous injection either once daily on Days 1 through 42, or twice weekly on Days 1 through 39 or once weekly on Days 1 through 36.

This single-center trial was conducted in the United States. The overall time to participate in this study is up to 56 days. Participants made daily visits to the clinic for 8 weeks, and were contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has total serum testosterone (ST) levels less than 300 ng/dL at Screening.
2. Has a body mass index (BMI) between 20.0 and 40.0 kg/m^2, inclusive at Screening.
3. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from the time of signing of informed consent throughout the duration of the study and for 12 weeks after the last dose.

Exclusion Criteria:

1. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality that may impact the ability of the participant to participate or potentially confound the study results. Participants will be excluded based on:

   1. Has a serum creatinine >2.0 milligrams per deciliter (mg/dL) at Screening.
   2. Is receiving dialysis treatment.
   3. Has an American Urological Association (AUA)/ International Prostate Symptom Score (I-PSS) score of >19 or serum prostate-specific antigen (PSA) >4 nanogram per milliliter (ng/mL) at Screening.
   4. Has thyrotropin (TSH) levels less than (<) 0.3 or >7.5 milli-international units per liter (mIU/L) at Screening.
   5. Has systolic blood pressure >160 millimeter of mercury (mm Hg) or diastolic blood pressure >100 mm Hg (if out of range may be repeated once for eligibility determination) at Screening.
   6. Has luteinizing hormone (LH) >9.4 units per liter (U/L) at Screening.
   7. Is receiving insulin therapy.
   8. Has a hematocrit <30 percent (%) or >48% at Screening.
   9. Has a glycosylated hemoglobin (HbA1c) >8.0 at Screening (Cohort 1).
2. Has type 2 diabetes mellitus defined as fasting blood glucose >125 mg/dL, glycosylated hemoglobin (HbA1c) >6.2%, or use of antidiabetic medication (Cohort 2 only).
3. Has clinical evidence of anatomic or pathological hypothalamic/pituitary/testicular disease, such as (but not limited to) Klinefelter's syndrome, Kallmann's syndrome, systemic infiltrative diseases (hemochromatosis, sarcoidosis, Wilson's disease), or prior pituitary surgery.
4. Has used gonadotropin-releasing hormone (GnRH) agonists, GnRH antagonists, antiandrogens, clomiphene, or other reproductive hormone-related agents within 6 months prior to Screening.
5. Has used anabolic therapies (testosterone, dehydroepiandrosterone [DHEA], androstendione, any other androgen, or recombinant human growth hormone) within 1 year of Screening.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 10 September 2015 to 08 April 2016.
Pre-assignment Details: Middle-aged and older male participants with low testosterone levels were enrolled in once daily TAK-448 0.1 µg, twice weekly TAK-448 0.3 µg, once weekly TAK-448 1 µg or Placebo groups.
Groups:
- TAK-448 0.1 µg: TAK-448 0.1 mcg, injection, subcutaneously, once daily on Days 1 through 42.
- TAK-448 0.3 µg: TAK-448 0.3 µg, injection, subcutaneously, twice-weekly on Days 1 through 39.
- TAK-448 1.0 µg: TAK-448 1.0 µg, injection, subcutaneously, once-weekly on Days 1 through 36.
Period: Overall Study
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Started | 5 | 2 | 5 | 5
Completed | 5 | 2 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Groups:
- TAK-448 0.1 µg: TAK-448 0.1 µg, injection, subcutaneously, once daily on Days 1 through 42.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg | Total
Number analyzed (Participants) | 5 | 2 | 5 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (3.24) | 71.0 (11.31) | 70.6 (9.32) | 65.2 (1.48) | 67.1 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 2 | 5 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic and Latino | 5 | 2 | 5 | 5 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 3 | 3
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 5 | 1 | 4 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 5 | 5 | 17
Height [Mean (Standard Deviation); unit: cm] | 173.6 (5.81) | 173.5 (3.54) | 172.4 (7.80) | 174.6 (6.77) | 173.5 (6.05)
Weight [Mean (Standard Deviation); unit: kg] | 93.0 (16.6) | 101.6 (11.3) | 99.4 (17.3) | 91.5 (21.5) | 95.5 (16.8)
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (4.3) | 33.9 (5.2) | 33.3 (4.2) | 30.0 (6.5) | 31.6 (4.9)
Smoking Classification [Number; unit: participants]
  Participant has never smoked | 3 | 1 | 3 | 4 | 11
  Participant is an ex-smoker | 2 | 1 | 2 | 1 | 6
Alcohol Classification [Number; unit: participants]
  Participant has never drunk | 1 | 1 | 0 | 0 | 2
  Participant is a current drinker | 3 | 1 | 3 | 5 | 12
  Participant is an ex-drinker | 1 | 0 | 2 | 0 | 3
Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 2 | 3 | 4 | 12
  No | 2 | 0 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Average Serum Concentration (Cav) of Total ST After 6 Weeks of Dosing
Description: Cav is the average serum concentration of the dosing interval, calculated as area under the effect curve (AUEC) divided by the duration of the dosing interval.
Time Frame: Once-daily regimen Day 42; Twice-weekly regimen Day 39; Once-weekly regimen Day 36
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug or placebo and who had at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 5 | 2 | 5 | 5
percent change | 14.32 (29.186) | 7.100 (18.102) | 10.60 (12.594) | 15.80 (26.531)

2. Primary Outcome: Trough Serum Concentration (Ctrough) of ST
Description: Trough serum concentration of total and free ST, defined as lowest Baseline concentration.
Time Frame: Once-daily regimen Day 42; Twice-weekly regimen Day 39; Once-weekly regimen Day 36
Population: PD analysis set included all participants who received at least 1 dose of study drug or placebo and who had at least 1 valid PD measure. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 5 | 2 | 4 | 5
ng/dL | 285.4 (94.952) | 255.5 (102.53) | 135.3 (44.515) | 244.4 (61.756)

3. Secondary Outcome: Serum Testosterone Cmax: Maximum Observed Plasma Concentration
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Assessments were done Day 1 and Day 42 for once daily regimen, on Day 36 for once weekly regimen and on Day 39 for twice-weekly regimen (Day 42/36/39).
Time Frame: Day 1 (first dose) and Day 42 for once-daily regimen, Day 39 for twice-weekly regimen, or Day 36 for once-weekly regimen (last dose)
Population: PD analysis set included all participants who received at least 1 dose of study drug or placebo and who have at least 1 valid PD measure.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 5 | 2 | 5 | 5
ng/dL
  Day 1 | 287.6 (58.518) | 306.5 (68.589) | 351.2 (87.434) | 427.8 (67.054)
  Day 42/36/39 | 354.8 (136.09) | 287.0 (57.983) | 263.8 (82.914) | 343.0 (57.524)

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for the Free Form of TAK-448 (TAK-448F)
Description: Cmax is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Once-daily Dosing Days 1 and 42, Twice-weekly Dosing Days 1 and 39, Once-weekly Dosing Days 1 and 36, predose and at multiple time intervals (up to 8 hours) post-dose.
Population: Due to early termination of the study pharmacokinetic data was not collected and reported.
Arm/Group | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: AUCt: Area Under the Plasma Concentration-Time Curve for TAK-448F
Description: Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Time Frame: as for outcome 4
Population: Due to early termination of the study pharmacokinetic data was not collected and reported.
Arm/Group | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Terminal Elimination Half-life (T1/2) for TAK-448F
Description: T1/2 is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 4
Population: Due to early termination of the study pharmacokinetic data was not collected and reported.
Arm/Group | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 56
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-448 0.1 µg | TAK-448 0.3 µg | TAK-448 1.0 µg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 1/2 | 4/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | TAK-448 0.1 µg (N=2) | TAK-448 0.3 µg (N=5) | TAK-448 1.0 µg (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.